CLINICAL TRIAL: NCT05286476
Title: Effect of 6 Weeks of Whole-body Vibration in Treatment of Postnatal Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohamed othman, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: /012/002926
Record Dates: First submitted 2022-02-28; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Constipation
Keywords: Whole Body Vibration; Postnatal women
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): received Whole-body Vibration, pelvic floor exercise and static abdominal exercises interventions In addition to diet instructions
  Interventions: Combination Product: Whole Body Vibration; Other: pelvic floor exercises and static abdominal exercises in addition to diet instructions
- group B (Other): received pelvic floor exercises and static abdominal exercises in addition to diet instructions only
  Interventions: Other: pelvic floor exercises and static abdominal exercises in addition to diet instructions

INTERVENTIONS:
Combination Product: Whole Body Vibration — vibration was administered for 1min, with a rest interval of 1min between each vibration set repeating 10 vibrations, with a frequency of 30 Hz and an amplitude of 0-2 mm and a speed of 50 m /s,18 and these sessions lasted for 6 weeks 3 days a week. whole-body vibration was induced by a noninvasive oscillation platform
  Other Names: pelvic floor exercises and static abdominal exercises in addition to diet instructions only
  Arms: group A
Other: pelvic floor exercises and static abdominal exercises in addition to diet instructions — During the low abdominal hollowing with instructed pelvic floor co-contraction test subjects were instructed with the standard command: 'Breathing normally, and keeping your back still, gently lift and tighten your pelvic floor. Now gently draw in your low tummy as well and hold it'. Pelvic floor facilitates transversus abdominis thickness.
  subject in supine lying with her arms crossed over the diastasis for support. And subject has to draw or pull the abdomen inwards so that there elicits an isometric contraction of abdominal muscles and repeated this for 5-7 times.

SUMMARY:
Background: Postpartum constipation is a common problem affecting postpartum mothers. Aim: To determine whether Whole Body Vibration is effective in treatment of postnatal women constipation. Design: The study was designed as a prospective, randomized, single-blind, pre-post-test, controlled trial.

HYPOTHESES:

It will be hypothesized that:

It was hypothesized that whole-body vibration has no or limited effect in treatment of postnatal constipation RESEARCH QUESTION: Does whole-body vibration has an effect in treatment of postnatal constipation?

DETAILED DESCRIPTION:
Methods: Group A received whole-body vibration, pelvic floor exercise and static abdominal exercises interventions for six weeks and group B received pelvic floor exercises and static abdominal exercises in addition to diet instructions in both groups. Constipation symptom questionnaire and patient assessment of constipation quality of life questionnaire is applied before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participants age ranged from 22 to 35 years old
* with vaginal delivery
* complain from postnatal constipation from (2 - 6 weeks) post-delivery
* had body mass index (BMI) ranged from 30 to 32 kg/m2.

Exclusion Criteria:

Participants were excluded if they:

* had diabetes, hypertension, cardiac diseases.
* Women who had history of inflammatory bowel disease and abnormalities of anal region or anal fissure
* women who had history of bowel surgery (other than appendectomy),
* patients who had endocrine disease or digestive tract disease
* history of neurological or musculoskeletal disorder.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females complains from postnatal constipation
Enrollment: 40 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Patient Assessment of Constipation-Symptom questionnaire | Change from Baseline then after 6 weeks of intervention.
  PAC-SYM is composed of three domains: abdominal symptoms, 4 items; rectal symptoms, 3 items; and stool symptoms, 5 items. Wording was as follows: ''How severe have each of these symptoms been in the last two weeks?'' Items are rated on a 5-point (0-4) Likert scale. Responses are scored as 0 = absence of symptom, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe. The ABD, REC and STO domain scores are the mean scores of each domain. Constipation was defined by the responses to the following questions: ''Have laxatives been taken during this period?'' (if ''yes'' then CC = 0: end of scoring); ''Have stools been passed on 3 or more days/week on average?'' (if ''yes'' then F = 0; if ''no'' then F = 1: in either case, and for subsequent questions, scoring is continued); ''Was stool passage difficult or painful?'' and ''Was stool consistency predominantly hard?'' The CC score indicates either constipation (CC = 2 or 3) or non-constipation (CC = 0 or 1).
Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) | Change from Baseline then after 6 weeks of intervention.
  PAC-QOL questionnaire comprises 28 questions and depending on the factor analysis structure, the tool comprises four subscales, including "Physical discomfort (question 1-4)," "Psychosocial discomfort (question 5-12)," "Worries and concerns (question 13-23)," and "Satisfaction (question 24-28)." Similar to the Likert scale, each option is scored on a scale of 0-4 (least to the greatest effect), and higher scores indicate a worst quality of life. However, reverse coding was required in questions 18, 25, 26, 27, and 28 because they were positive questions, whereas the other 23 questions were negative ones.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa raafat, PhD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in bee venom or ulcer . we will share the results of this study within 1 year following publication
Supporting Information: SAP, ICF
Time Frame: 1 year after publication
Access Criteria: the criteria will be assessed by the publication of the trial in an international journals.

REFERENCES:
- [Derived] Elfatah Elhosary EA, ElAzab DR, Hanoura EM, Othman EM. Effect Of Six Weeks Of Whole-Body Vibration In Treatment Of Postnatal Constipation. J Pak Med Assoc. 2023 Apr;73(Suppl 4)(4):S13-S16. doi: 10.47391/JPMA.EGY-S4-3. PMID 37482821